Study Protocol and Statistical Analysis Plan

Brief Title: Correlation Between Carotid Stump Pressure and Interhemispheric rSO<sub>2</sub>

Asymmetry During Awake Carotid Endarterectomy

Official Title: Evaluation of the Correlation Between Carotid Stump Pressure and

Interhemispheric rSO<sub>2</sub> Asymmetry in Awake Carotid Endarterectomy: A Prospective Cohort

Study

Document Date: August 2025

NCT Number: [to be assigned upon registration]

Background and Rationale

Carotid artery stenosis accounts for 15-30% of ischemic strokes. Carotid

endarterectomy (CEA) reduces recurrent stroke risk in patients with significant stenosis but

carries intraoperative risk of cerebral hypoperfusion during carotid cross-clamping. Carotid

stump pressure (SP) is used as a surrogate for collateral circulation, while near-infrared

spectroscopy (NIRS) provides a continuous, non-invasive estimate of regional cerebral oxygen

saturation (rSO<sub>2</sub>). Limitations exist with both, and no universal threshold has been validated.

Recent interest has shifted toward interhemispheric rSO<sub>2</sub> asymmetry as a marker of perfusion

adequacy with different clinical conditions. This study investigates whether SP differs

significantly between patients with asymmetry >10% and those with asymmetry ≤10%

Study Objectives

Primary Objective

To determine whether stump pressure values differ significantly between patients with

interhemispheric rSO<sub>2</sub> asymmetry >10% vs. ≤10% during awake CEA.

Secondary Objectives

1. Interhemispheric asymmetry difference.

2. Assess correlation between SP and interhemispheric  $\Delta rSO_2$  difference.

3. Assess correlation between SP and ipsilateral  $\Delta rSO_2$ .

4. Identify a carotid SP threshold predictive of significant asymmetry using ROC curve

analysis.

5. Evaluate the independent predictive value of SP for asymmetry using multivariable

logistic regression (adjusted for age, sex, carotid stenosis, intraoperative

hemodynamics).

6. Compare intraoperative hemodynamic parameters (PaO<sub>2</sub> (partial pressure of arterial

oxygen), SpO<sub>2</sub> (peripheric oxygen saturation), systolic blood pressure, heart rate) and

procedural variables (need for shunt, cross-clamp duration, surgical time) between

groups.

7. Document postoperative complications (neurological deficit, bleeding) within 30 days.

Study Design

Type: Single-center, prospective observational cohort study

Setting: Tertiary academic hospital (Cardiovascular Surgery Department)

Population: Adult patients undergoing elective awake CEA under regional anesthesia (superficial cervical plexus block)

Sample Size: ~60 patients (based on power analysis)

## Groups:

Asymmetry group: >10% interhemispheric ΔrSO<sub>2</sub> difference

Symmetry group: ≤10% interhemispheric ΔrSO₂ difference

Time Perspective: Prospective, 30 days.

Masking: None (open-label observational study)

## Eligibility Criteria

## Inclusion Criteria:

- 1. Age ≥18 years
- 2. Elective CEA under regional (superficial cervical plexus block) anesthesia
- 3. Bilateral rSO<sub>2</sub> monitoring with NIRS
- 4. Successful SP measurement after cross-clamping
- 5. Written informed consent

## **Exclusion Criteria:**

- 1. Incomplete SP or NIRS data
- 2. Conversion to general anesthesia
- 3. Intraoperative technical complications
- 4. Prior ipsilateral CEA or stenting
- 5. Major disabling stroke
- 6. MI within 3 months
- 7. Traumatic brain injury within 6 months

**Intervention and Monitoring** 

Anesthesia: Superficial cervical plexus block.

Monitoring: ECG, SpO<sub>2</sub>, invasive arterial pressure, bilateral frontal NIRS (INVOS 5100C).

Procedure: Standard CEA under regional anesthesia; SP measured 3 min after cross-clamping

with 22G catheter.

**Data Collection Points:** 

T1: Baseline (before cross-clamping)

T2: 3 minutes after cross-clamp

**Outcome Measures** 

Primary Outcome:

Difference in carotid stump pressure between asymmetry (>10% ΔrSO<sub>2</sub>) and symmetry  $(\leq 10\% \Delta rSO_2)$  groups.

Time frame: 3 minutes post-cross-clamp.

**Secondary Outcomes:** 

- 1. Interhemispheric asymmetry difference.
- 2. Correlation between SP and interhemispheric ΔrSO<sub>2</sub> difference (3 min post-clamp).
- 3. Correlation between SP and ipsilateral  $\Delta rSO_2$  (3 min post-clamp).
- 4. ROC curve threshold analysis for SP predicting asymmetry.
- 5. Logistic regression model (SP + covariates).
- 6. Comparison of intraoperative hemodynamics and procedural characteristics between groups.

7. Postoperative neurological or bleeding complications within 30 days.

Statistical Analysis Plan

Descriptive statistics: Continuous data as mean  $\pm$  SD or median (IQR); categorical as frequency/%.

Normality test: Shapiro-Wilk.

Primary outcome: Independent t-test (SP difference between groups). Mann–Whitney U if non-parametric.

Secondary outcomes:

Spearman's correlation (SP vs.  $\Delta rSO_2$ , ipsilateral  $\Delta rSO_2$ ).

ROC analysis to determine SP cutoff for asymmetry (>10%).

Logistic regression (Model 1: SP; Model 2: adjusted for age, sex, stenosis; Model 3: + intraoperative variables).

Hemodynamic/procedural comparisons: t-test, Mann-Whitney, or Fisher's exact test.

30-day complications compared between groups (Fisher's exact).

Significance threshold: p < 0.05.

Software: IBM SPSS v26.

Power Analysis

Preliminary data:

Symmetry group SP:  $56 \pm 15$  mmHg

Asymmetry group SP:  $44 \pm 13$  mmHg

Cohen's d = 0.855

Sample size calculation (two-sample t-test,  $\alpha = 0.05$ , power = 0.90, two-tailed):

Required per group =  $\sim 30$  patients

Total =  $\sim$ 60 patients

Software: G\*Power 3.1

Ethics

Approval: Izmir Katip Celebi University Health Research Ethics Committee

Approval No: 0442 (17 July 2025)

Conducted per the Declaration of Helsinki.

Written informed consent required.

**Data Sharing** 

Plan: De-identified IPD (SP values, rSO<sub>2</sub> data, intraoperative hemodynamics, outcomes) will be available upon reasonable request for academic purposes.

Access: Requests subject to institutional and ethical approval.